CLINICAL TRIAL: NCT06135870
Title: Role of Senescent Cells in Uterine Fibroid Pathogenesis
Brief Title: Role of Senescent Cells in Uterine Fibroid Pathogenesis (SOUL Study)
Acronym: SOUL
Status: Recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00359032; 1R01HD111243 (NIH)
Record Dates: First submitted 2023-11-09; First posted 2023-11-18 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Fibroid; Leiomyoma
Keywords: Senescent cells; Fibroids; Leiomyomas
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fibroid, myometrial samples, and peripheral blood sample.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with fibroids undergoing elective hysterectomy or myomectomy: Women between the age of 18-55 with fibroids undergoing elective hysterectomy or myomectomy

SUMMARY:
The investigators are evaluating the role of senescent cells in uterine fibroids.

DETAILED DESCRIPTION:
Uterine fibroids are prevalent tumors of uterus characterized by excessive fibrotic tissues. Using new cutting-edge computational methods, the investigators have found that small groups of senescent cells in fibroids work in concert with immune cells to produce soluble factors in fibroid tissues to create a feed-forward loop leading to fibrosis. This project seeks to unravel key cell-cell communication networks involving senescent and immune cells in fibroids to develop new treatments for uterine fibroids.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be women above the age of ≥18 - ≤55 years.
* Women with suspected uterine fibroids.
* Subject must be or have been sexually active or have had a previous vaginal exam that used a speculum.
* Subject must be able to understand, read and speak English or Spanish and subsequently, be able to understand what she is consenting to in terms of procedures and use/disclosure of protected health information.

Exclusion Criteria:

* Unwilling to sign the consent form or complete questionnaire.
* Pregnancy.
* Cancer of the uterus

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women between the age of 18-55 years undergoing elective hysterectomy or myomectomy for uterine fibroids
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Develop an atlas to comprehensively quantify the rate of senescent cell (SnC) types in fibroid and myometrium tissue samples | 5 years
  Perform scRNASeq on human fibroids and control myometrium tissue and apply transfer learning algorithm for SnC identification and phenotyping to identify cell-cell communication patterns in fibroids versus control myometrial tissue using Domino to validate computationally predicted senescent cell types. The computationally predicted immune phenotypes will be validated with flow cytometry.

SECONDARY OUTCOMES:
Validate the concentration senescence-associated secretory profile (SASP) in cell cultures of senescent cells in uterine fibroids | 5 years
  Quantify levels of transcripts and proteins in the fibroid senescence-associated secretory profile (SASP) using ELISA and western blotting techniques
Rate of inhibition of cellular proliferation and ECM deposition by senolytics and senomorphics in fibroids | 5 years
  Examine the in-vitro effects of senotherapeutcis using leiomyoma culture models and in mouse models. Measured by inhibition of proliferation, induction of apoptosis, inhibition ECM deposition, decrease in SnCs (senolytics) and senescence-associated secretory profile SASPs (senomorphics).

CONTACTS AND LOCATIONS:
Overall Officials: James Segars, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No